CLINICAL TRIAL: NCT04198103
Title: Transperineal Laser Ablation for Percutaneous Treatment of Benign Prostatic Hyperplasia: A Feasibility Study - Results at 6 and 12 Months From a Retrospective Multi-centric Study
Brief Title: Transperineal Laser Ablation for Percutaneous Treatment of Benign Prostatic Hyperplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Rome Tor Vergata (Other)
Collaborators: Ospedale Regina Apostolorum (Other); European Institute of Oncology (Other)
Responsible Party: Principal Investigator, Guglielmo Manenti, Principle Investigator, University of Rome Tor Vergata
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS.99
Record Dates: First submitted 2019-11-08; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: BPH; Lower Urinary Tract Symptoms
Keywords: BPH; LUTS
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SoracteLite (Experimental): Transperineal Focal Laser Ablation (TPLA)
  Interventions: Device: Transperineal Focal Laser Ablation (TPLA)

INTERVENTIONS:
Device: Transperineal Focal Laser Ablation (TPLA) — The intervention will take place in an ambulatory setting using EchoLaser system. The treatment consists of the trasmission of laser energy into the tissue through the percutaneous insertion of optical fiber under local anesthesia. Within each needle, an optic fiber of 300 µm will be inserted. Each ablation lasts 6 minutes and each fiber ablates 1800J at a power of 3W. At the end of the first ablation there is a pull-back of about 1 cm from the original ablation location. According to the dimension of the middle lobe of the prostate, multiple pullbacks can be used for a total duration of about 30minutes. At the end of the treatment corticosteroid is given for anti-edema and anti-inflammatory effects and Antibiotic therapy and gastroprotective therapy is given. After an adequate amount of time for observation, the patient is dismissed.
  Other Names: SoracteLite EchoLaser

SUMMARY:
This study investigated the effectiveness and safety of SoracteLite ™- Trans-Perineal Laser ablation (TPLA) in the treatment of patients with symptomatic Benign Prostatic Hyperplasia (BPH) at 6 and 12 months follow-up

DETAILED DESCRIPTION:
The purpose of this study was to investigate the effectiveness and safety of SoracteLite ™ - Trans-Perineal Laser ablation (TPLA) in the treatment of patients with symptomatic benign prostatic hyperplasia (BPH) at 6 and 12 months follow-up. Methods: Patients with urinary symptoms secondary to BPH underwent TPLA under local anaesthesia in four centers. Under US guidance, up to four 21G applicators were inserted in the prostatic tissue. Each treatment was performed with diode laser operating at 1064 nm changing the illumination time according to prostate size.

ELIGIBILITY:
Inclusion Criteria:

* Male
* ≥ 50 years of age
* International Prostate Symptoms (IPSS) ≥12
* Peak urinary flow rate (Qmax): <15 ml
* Prostate volume: ≥ 30 ml, measured by transrectal ultrasound
* Post-void residual (PVR): <400 ml
* Signed informed consent

Exclusion Criteria:

* MRI signs of malignancy confirmed by biopsy investigation
* urethral stenosis
* serious coagulation disorders
* inadequate compliance
* ischemic pathology in the previous six months
* active phase inflammatory pathology

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical symptoms changes at 6 months and 12 months follow-up evaluated with objective and subjective parameters | 12 months
  Improvement of obstructive symptomatology correlated to BPH. The evaluation will be based on urodynamic studies of Qmax, post void and residual volume

SECONDARY OUTCOMES:
Treatment safety measured by complications incidence | 30 days
  Number of incidence of Complication according to modified Clavien classification system

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Casa di Cura Santa Rita, Atripalda, AV
  - ASST Bergamo Est, Seriate, BG
  - Policlinico Tor Vergata (PTV) Foundation: UOC Department of Diagnostic Imaging and Interventional Radiology, Rome, RM
  - IGreco Ospedali Riuniti, Cosenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patelli G, Ranieri A, Paganelli A, Mauri G, Pacella CM. Transperineal Laser Ablation for Percutaneous Treatment of Benign Prostatic Hyperplasia: A Feasibility Study. Cardiovasc Intervent Radiol. 2017 Sep;40(9):1440-1446. doi: 10.1007/s00270-017-1662-9. Epub 2017 May 4. PMID 28474112
- [Background] Raz O, Haider MA, Davidson SR, Lindner U, Hlasny E, Weersink R, Gertner MR, Kucharczyk W, McCluskey SA, Trachtenberg J. Real-time magnetic resonance imaging-guided focal laser therapy in patients with low-risk prostate cancer. Eur Urol. 2010 Jul;58(1):173-7. doi: 10.1016/j.eururo.2010.03.006. Epub 2010 Mar 12. PMID 20334965
- [Background] Lindner U, Weersink RA, Haider MA, Gertner MR, Davidson SR, Atri M, Wilson BC, Fenster A, Trachtenberg J. Image guided photothermal focal therapy for localized prostate cancer: phase I trial. J Urol. 2009 Oct;182(4):1371-7. doi: 10.1016/j.juro.2009.06.035. Epub 2009 Aug 14. PMID 19683262
- [Background] Goldberg SN, Grassi CJ, Cardella JF, Charboneau JW, Dodd GD 3rd, Dupuy DE, Gervais D, Gillams AR, Kane RA, Lee FT Jr, Livraghi T, McGahan J, Phillips DA, Rhim H, Silverman SG; Society of Interventional Radiology Technology Assessment Committee. Image-guided tumor ablation: standardization of terminology and reporting criteria. J Vasc Interv Radiol. 2005 Jun;16(6):765-78. doi: 10.1097/01.RVI.0000170858.46668.65. PMID 15947040
- [Background] Bremer C, Kreft G, Roggan A, Filler T, Reimer P. Ex vivo evaluation of novel miniaturized laser-induced interstitial thermotherapy applicators for effective small-volume tissue ablation. Invest Radiol. 2001 Jun;36(6):327-34. doi: 10.1097/00004424-200106000-00005. PMID 11410753
- [Background] Costello AJ, Bowsher WG, Bolton DM, Braslis KG, Burt J. Laser ablation of the prostate in patients with benign prostatic hypertrophy. Br J Urol. 1992 Jun;69(6):603-8. doi: 10.1111/j.1464-410x.1992.tb15631.x. PMID 1379101